CLINICAL TRIAL: NCT07251686
Title: Impact of Extubation Technique on Postoperative Pulmonary Outcomes: A Randomized Controlled Trial
Brief Title: Positive-Pressure vs Suction Extubation in Cesarean Patients
Acronym: PPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, NURDAN YILMAZ, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPETRCT2024; Medipol University Ethics (Other: Ethics Approval No: 2025/1065(Medipol University))
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Respiratory Complication; Atelectasis; Anesthesia, General; Extubation; Hypoxia
Keywords: Postoperative Respiratory Complication; Positive pressure; Extubation; Cesarean Section; Anesthesia; Hypoxia
MeSH Terms: conditions — Pulmonary Atelectasis; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded because all procedures were performed under general anesthesia, and they were unaware of which extubation technique was used. The anesthesiologist performing extubation was not blinded to group allocation. Postoperative oxygenation data were recorded and analyzed by an investigator blinded to the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive-Pressure Extubation (PPET) (Experimental): Extubation was performed under continuous positive airway pressure (PEEP 6 cmH₂O, PS 12 cmH₂O) during cuff deflation.
  Interventions: Procedure: Positive Pressure Extubation Technique (PPET)
- Negative-Pressure Extubation (NPET) (Active Comparator): Extubation was performed under continuous suction during cuff deflation, representing the conventional technique.
  Interventions: Procedure: Negative Pressure Extubation Technique (NPET)

INTERVENTIONS:
Procedure: Negative Pressure Extubation Technique (NPET) — Extubation performed under continuous suction during cuff deflation.
  Arms: Negative-Pressure Extubation (NPET)
Procedure: Positive Pressure Extubation Technique (PPET) — Extubation performed under continuous positive airway pressure during cuff deflation (PEEP 6 cmH₂O, PS 12 cmH₂O)
  Arms: Positive-Pressure Extubation (PPET)

SUMMARY:
This randomized controlled trial aims to evaluate the effects of two tracheal extubation techniques on postoperative oxygenation and early respiratory outcomes in adult women undergoing elective cesarean delivery under general anesthesia. A total of 120 participants will be randomly assigned to the Positive Pressure Extubation Technique (PPET) group or the Negative Pressure Extubation Technique (NPET) group.

In the PPET group, extubation will be performed while maintaining positive airway pressure during cuff deflation, whereas in the NPET group, extubation will be performed under continuous suction. The primary outcome will be the incidence of postoperative desaturation, defined as peripheral oxygen saturation (SpO₂) below 92% within the first 60 minutes after extubation.

Secondary outcomes will include serial measurements of oxygen saturation, heart rate, and blood pressure, along with exploratory analyses assessing the relationship between body mass index, comorbidities, and desaturation risk. The trial is intended to determine whether PPET provides physiological advantages over NPET during tracheal extubation in this surgical population.

DETAILED DESCRIPTION:
Extubation represents a vulnerable phase of general anesthesia, during which airway secretions, reduced functional residual capacity, and diminished upper airway tone may contribute to hypoxemia and other respiratory complications. Pregnant women are particularly susceptible due to decreased lung volumes, increased oxygen consumption, and airway edema associated with pregnancy.

The Positive-Pressure Extubation Technique (PPET) has been proposed as a strategy to reduce the migration of secretions toward the distal airways during cuff deflation, potentially improving lung aeration and gas exchange. Unlike conventional suction-based methods, PPET uses continuous positive pressure to maintain airflow direction, theoretically minimizing micro-aspiration and early atelectasis formation.

Although PPET has demonstrated benefits in pediatric and mixed surgical populations, evidence regarding its application in obstetric anesthesia remains scarce. This study aims to evaluate whether positive-pressure extubation provides physiological advantages over conventional negative-pressure extubation in adult patients undergoing cesarean delivery under general anesthesia. By examining postoperative respiratory stability and hemodynamic responses, the study is expected to clarify the clinical importance of tailored extubation strategies in populations with reduced pulmonary reserve.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients aged 18 to 45 years.
* Scheduled for elective cesarean delivery under general anesthesia.
* Ability to provide written informed consent

Exclusion Criteria:

* Exclusion criteria included patients participating in another study,
* Patients refusing to participate,
* Uncooperative patients,
* Patients undergoing emergency surgery,
* American Society of Anesthesiologists (ASA) Physical Status Classification > 3,
* Patients with chronic respiratory failure, obstructive sleep apnea, and patients with anticipated difficult airways.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only adult female patients undergoing elective cesarean section under general anesthesia were enrolled.
Enrollment: 120 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative desaturation (SpO₂ < 92%) | Within the first 60 minutes after extubation
  The proportion of participants who experience oxygen desaturation, defined as peripheral oxygen saturation (SpO₂) below 92%, at any time point within the first 60 minutes after extubation.

SECONDARY OUTCOMES:
Change in Peripheral Oxygen Saturation (SpO₂) | 0-60 minutes post-extubation
  SpO₂ values measured at predefined intervals (1, 3, 5, 10, 15, 30, and 60 minutes) after extubation.
Change in Heart Rate | 0-60 minutes post-extubation
  Heart rate measurements recorded at predefined intervals after extubation.
Change in Systolic and Diastolic Blood Pressure | 0-60 minutes post-extubation
  Systolic and diastolic blood pressure were recorded at predefined intervals after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: NURDAN YILMAZ, Principal Investigator — Istanbul Medipol Mega University Hospital
Locations (1):
- Istanbul Medipol Mega University Hospital, Istanbul, Bagcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient confidentiality and institutional policy. Summary data will be available upon reasonable request from the corresponding author.